CLINICAL TRIAL: NCT01759342
Title: The Efficacy of a Standardized Exercise Protocol in Inpatient Care of Patients With Cystic Fibrosis
Brief Title: Comprehensive Exercise Training Program During Hospitalization for an Acute CF Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12.21.2012
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2012-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; pulmonary exacerbation, exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise; Resistance Training; Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive exercise program (Experimental): Moderate to high intensity aerobic, resistance, flexibility, posture and balance exercise program
  Interventions: Behavioral: Aerobic exercise; Behavioral: Resistance exercise; Behavioral: Flexibility and postural exercise; Behavioral: Balance exercise
- Usual care exercise (Active Comparator): 30 minutes/day of self selected mode and intensity of aerobic exercise
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise
Behavioral: Resistance exercise
  Arms: Comprehensive exercise program
Behavioral: Flexibility and postural exercise
  Arms: Comprehensive exercise program
Behavioral: Balance exercise
  Arms: Comprehensive exercise program

SUMMARY:
This protocol was designed to assess if when subjects with CF are admitted to the hospital for a pulmonary exacerbation if a comprehensive exercise program (moderate to high intensity aerobic, resistance, flexibility and balance exercises) was superior to our "usual care intervention (30 min/day of self selected mode and intensity of exercise) in improving aerobic capacity, muscle strength/power, flexibility and balance.

DETAILED DESCRIPTION:
This protocol was designed to assess if when subjects with CF are admitted to the hospital for a pulmonary exacerbation if a comprehensive exercise program (moderate to high intensity aerobic, resistance, flexibility and balance exercises) was superior to our "usual care intervention (30 min/day of self selected mode and intensity of exercise) in improving aerobic capacity, muscle strength/power, flexibility and balance.

The experimental group will participate in the following regime:

Day 1 - Evaluation including standardized tests and measures: If Day 1 is a M,W, F, day 2 will constitute: aerobic exercise between 20-30 minutes based on patient tolerance using the appropriate RPE scale (13-15 on Borg with patients ages 13-21, and 6-8 on pictoral CERT with patients ages 6-12)to ensure correct intensity. Choices will include treadmill, stationary bike, game bike, or ambulating at varying intensities throughout hospital; Balance Activities: Standing on bosu ball while performing UE activity (throwing, catching with another ball, Frisbee, etc.). Standing on one leg or B LE's will be determined by patients currently level.

If Day 1 is a Tuesday or Thursday, day 2 will constitute: 5-10 minutes of aerobic activity at warm up level (11-13 on Borg, and 4-6 on PCERT)x resistance training for UE: biceps, triceps, lattisimus, rhomboids/mid-trap, thoracic expansion exercises, and other muscles based on patient needs; resistance training for LE: quadriceps, hamstrings, gluteals (especially maximus and medius), and other muscles depending on patient need, core and abdominal strengthening, Stretches for flexibility depending on the patients individual needs: Thoracic expansion stretches will be done with every pt. supine and sidelying. Stretches are held for 10 seconds and repeated 10 times, Hamstring stretches will be performed if pt unable to reach line with sit and reach test.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 21 years
* admission for an acute Cystic fibrosis (CF) exacerbation
* forced expiratory volume in 1 s (FEV1) of < 60% of predicted at admission

Exclusion Criteria:

* medically unstable as deemed by the attending physician
* had completed both arms of the present study

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity following intervention of a comprehensive excercise training program | Participants will be followed for the duration of hospital stay, average number of days 10 (range 4 - 20 days)

SECONDARY OUTCOMES:
Muscle strength and power following intervention of a comprehensive excercise training program | Participants will be followed for the duration of hospital stay, average number of days 10 (range 4 - 20 days)
  Assessed with arm curl test, partial curl up test, timed 10 repetition sit to stand test
Posture/flexibility following intervention of a comprehensive excercise training program | Participants will be followed for the duration of hospital stay, average number of days 10 (range 4 - 20 days)
  Assessed with humeral distance, shoulder flexion range of motion, and hamstring length
Balance following intervention of a comprehensive excercise training program | Participants will be followed for the duration of hospital stay, average number of days 10 (range 4 - 20 days)
  Assessed with the pediatric Berg balance scale

CONTACTS AND LOCATIONS:
Overall Officials: John D Lowman, PT, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmimgham, Birmingham, Alabama, United States